CLINICAL TRIAL: NCT01054222
Title: A Local, Multicentre, Open-Label, Extension Trial To Evaluate The Efficacy And Safety Of Fesoterodine Flexible Dose Regimen In Elderly Patients With Overactive Bladder
Brief Title: Local, Open-Label, Extension Trial Of The Efficacy And Safety Of Fesoterodine In Elderly Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0221090
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-02

CONDITIONS: Urinary Bladder, Overactive
Keywords: overactive bladder idiopathic; elderly fesoterodine SOFIA Portugal extension study
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fesoterodine 4 mg (Other): Dose determined as per previous drug regime in A0221045 and investigator's evaluation.
  Interventions: Drug: Fesoterodine
- Fesoterodine 8 mg (Other): Dose determined as per previous drug regime in A0221045 and investigator's evaluation.
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine fumarate, sustained release (SR) tablet, 4 mg once daily, oral, duration - until fesoterodine is commercially available in Portugal or until 31 Dec 2011 (whichever is earlier)
  Other Names: Toviaz
  Arms: Fesoterodine 4 mg
Drug: Fesoterodine — Fesoterodine fumarate, sustained release (SR) tablet, 8 mg once daily, oral, duration - until fesoterodine is commercially available in Portugal or until 31 Dec 2011 (whichever is earlier)
  Other Names: Toviaz
  Arms: Fesoterodine 8 mg

SUMMARY:
This is an open-label extension study intended for subjects who have previously completed study A0221045 (fesoterodine in elderly OAB patients) and who have been recommended by the investigator as being suitable for the extended use of Fesoterodine. Data from this study will extend the evaluation of efficacy, tolerability and safety of Fesoterodine in older subjects from Portugal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have previously completed fesoterodine study A0221045 [in Portugal]
* Subjects must be recommended for inclusion by the investigator

Exclusion Criteria:

* Conditions or states excluding use of fesoterodine e.g. contraindication to fesoterodine
* Predominant stress incontinence as determined by the investigator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Portugal (3):
  - Centro de Avaliação Geriátrica, Lisbon
  - Hospital Ordem do Carmo, Porto
  - Hospital de São João, Porto

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221090&StudyName=Local%2C%20Open-Label%2C%20Extension%20Trial%20Of%20The%20Efficacy%20And%20Safety%20Of%20Fesoterodine%20In%20Elderly%20Patients%20With%20Overactive%20Bladder

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed treatment in study A0221045 (NCT00798434) were included in this study as per investigator's discretion.
Groups:
- Fesoterodine: Fesoterodine 4 milligram (mg) or 8 mg tablet orally once daily according to previous regime received in study A0221045 (NCT00798434).
Period: Overall Study
Arm/Group | Fesoterodine
Started | 31
Completed | 20
Not Completed | 11
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Fesoterodine
Number analyzed (Participants) | 31
Age Continuous [Mean (Standard Deviation); unit: Years] | 75.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Micturition-Related Urgency Episodes Per 24 Hours (End of Treatment [EOT])
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with Urinary Sensation Scale (USS) rating of greater than or equal to (>=) 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: End of Treatment (up to Week 82)
Population: Full analysis set (FAS): included all enrolled participants who had taken at least one dose of study treatment during the study and completed at least one micturition diary. Missing values were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
episodes per 24 hours | 5.48 (6.01)

2. Secondary Outcome: Mean Number of Micturition-Related Urgency Episodes Per 24 Hours
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18
Population: Full analysis set (FAS): included all enrolled participants who had taken at least one dose of study treatment during the study and completed at least one micturition diary. 'n' signifies participants who were evaluable for this measure at specified time points. Missing values were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
episodes per 24 hours
  Baseline (n= 28) | 10.49 (5.28)
  Month 3 (n= 25) | 5.28 (7.33)
  Month 6 (n= 28) | 6.37 (6.74)
  Month 9 (n= 28) | 4.98 (6.41)
  Month 12 (n= 28) | 5.15 (6.62)
  Month 15 (n= 27) | 5.09 (6.46)
  Month 18 (n= 24) | 5.22 (6.18)

3. Secondary Outcome: Mean Number of Severe Micturition-Related Urgency Episodes Per 24 Hours
Description: The mean number of severe micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to (>=) 4 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
episodes per 24 hours
  Baseline (n= 28) | 6.35 (6.90)
  Month 3 (n= 25) | 3.36 (7.14)
  Month 6 (n= 28) | 2.40 (6.15)
  Month 9 (n= 28) | 2.52 (5.84)
  Month 12 (n= 28) | 2.23 (5.86)
  Month 15 (n= 27) | 2.67 (6.08)
  Month 18 (n= 24) | 2.44 (6.27)
  End of Treatment (n= 28) | 2.29 (5.83)

4. Secondary Outcome: Mean Number of Micturitions Per 24 Hours
Description: Micturitions include episodes of voluntary micturition and episodes of Urgency Urinary Incontinence (UUI). UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
micturitions per 24 hours
  Baseline (n= 28) | 13.44 (4.57)
  Month 3 (n= 25) | 10.97 (4.72)
  Month 6 (n= 28) | 10.98 (4.26)
  Month 9 (n= 28) | 10.44 (4.26)
  Month 12 (n= 28) | 10.51 (4.46)
  Month 15 (n= 27) | 10.67 (4.06)
  Month 18 (n= 24) | 10.60 (4.41)
  End of Treatment (n= 28) | 10.38 (4.19)

5. Secondary Outcome: Mean Number of Nocturnal Micturitions Per 24 Hours
Description: Nocturnal micturitions were defined as micturitions with USS rating 1-5 that occurred between the time the participant went to bed and the time he or she arose to start the next day. USS rating: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. The mean number of nocturnal micturitions per 24 hours was calculated as the total number of nocturnal micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
micturitions per 24 hours
  Baseline (n= 28) | 3.45 (1.53)
  Month 3 (n= 25) | 3.08 (1.92)
  Month 6 (n= 28) | 3.25 (1.72)
  Month 9 (n= 28) | 3.07 (1.91)
  Month 12 (n= 28) | 2.88 (1.99)
  Month 15 (n= 27) | 3.00 (2.00)
  Month 18 (n= 24) | 2.95 (2.05)
  End of Treatment (n= 28) | 2.95 (2.05)

6. Secondary Outcome: Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours
Description: UUI episodes were defined as those with the USS rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
episodes per 24 hours
  Baseline (n= 28) | 2.64 (5.31)
  Month 3 (n= 25) | 2.27 (6.86)
  Month 6 (n= 28) | 1.54 (5.76)
  Month 9 (n= 28) | 1.36 (5.62)
  Month 12 (n= 28) | 1.29 (5.69)
  Month 15 (n= 27) | 1.83 (5.99)
  Month 18 (n= 24) | 1.65 (6.06)
  End of Treatment (n= 28) | 1.49 (5.62)

7. Secondary Outcome: Daily Sum Rating on the Urinary Sensation Scale (USS)
Description: The daily sum rating was calculated as the mean rating score on the USS multiplied by the mean number of micturitions per 24 hours at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine. Numerical decrease indicates improvement.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
Units on a Scale
  Baseline (n= 28) | 45.63 (23.72)
  Month 3 (n= 25) | 31.60 (30.32)
  Month 6 (n= 28) | 31.39 (26.10)
  Month 9 (n= 28) | 28.29 (25.75)
  Month 12 (n= 28) | 27.63 (26.66)
  Month 15 (n= 27) | 28.67 (26.31)
  Month 18 (n= 24) | 29.01 (26.87)
  End of Treatment (n= 28) | 28.60 (25.16)

8. Secondary Outcome: Percentage of Incontinent Participants at Baseline
Description: UUI episodes were defined as those with the urinary sensation scale (USS) rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline
Population: Full analysis set (FAS): included all enrolled participants who had taken at least one dose of study treatment during the study and completed at least one micturition diary.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 31
Percentage of Participants | 58.1

9. Secondary Outcome: Percentage of Participants With No Urgency Urinary Incontinence (UUI) Episode
Description: as for outcome 8
Time Frame: Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: FAS: all enrolled participants who had taken at least one dose of study treatment during study and completed at least one micturition diary. N (number of participants analyzed) signifies participants who had baseline UUI episodes >0 per 24 hours. 'n' signifies participants evaluable for this measure at specified time points. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 18
Percentage of Participants
  Month 3 (n= 16) | 81.3
  Month 6 (n= 18) | 77.8
  Month 9 (n= 18) | 77.8
  Month 12 (n= 18) | 77.8
  Month 15 (n= 17) | 64.7
  Month 18 (n= 15) | 66.7
  End of Treatment (n= 18) | 66.7

10. Secondary Outcome: Mean Number of Urinary Incontinence Pads, Barrier Creams and Powder Used Per 24 Hours
Description: The mean number of urinary incontinence pads (IP), barrier creams (BC) and powder used per 24 hours is calculated as the total number of IP, BC and powder used divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units per 24 hours
Arm/Group | Fesoterodine
Number analyzed (Participants) | 18
Units per 24 hours
  Baseline: IP (n= 18) | 3.69 (2.71)
  Baseline: BC (n= 18) | 0.48 (0.90)
  Baseline: Powder (n= 18) | 0.24 (1.02)
  Month 3: IP (n= 16) | 3.15 (4.63)
  Month 3: BC (n= 16) | 0.79 (2.07)
  Month 3: Powder (n= 16) | 0.19 (0.75)
  Month 6: IP (n= 18) | 3.02 (4.26)
  Month 6: BC (n= 18) | 0.43 (1.01)
  Month 6: Powder (n= 18) | 0.20 (0.86)
  Month 9: IP (n= 18) | 2.56 (2.34)
  Month 9: BC (n= 18) | 0.33 (1.07)
  Month 9: Powder (n= 18) | 0.17 (0.71)
  Month 12: IP (n= 18) | 2.52 (2.44)
  Month 12: BC (n= 18) | 0.13 (0.55)
  Month 12: Powder (n= 18) | 0.31 (1.34)
  Month 15: IP (n= 17) | 2.45 (2.32)
  Month 15: BC (n= 17) | 0.18 (0.53)
  Month 15: Powder (n= 17) | 0.00 (0.00)
  Month 18: IP (n= 15) | 2.49 (2.22)
  Month 18: BC (n= 15) | 0.18 (0.53)
  Month 18: Powder (n= 15) | 0.00 (0.00)
  End of Treatment: IP (n= 18) | 2.31 (2.11)
  End of Treatment: BC (n= 18) | 0.15 (0.49)
  End of Treatment: Powder (n= 18) | 0.00 (0.00)

11. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Month 3,6,9,12,15,18, and End of Treatment
Description: PPBC: self-administered, single-item, questionnaire that asked participants to describe their perception of their bladder-related problems. PPBC assessment rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Change = observation minus baseline. Results categorized as Deterioration (score difference ≥1), No Change (score difference=0), Improvement (score difference less than [<]0).
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
Participants
  Baseline: No Problems at all (n= 28) | 0
  Baseline: Some Very Minor Problems (n= 28) | 2
  Baseline: Some Minor Problems (n= 28) | 11
  Baseline: Some Moderate Problems (n= 28) | 11
  Baseline: Severe Problems (n= 28) | 4
  Baseline: Many Severe Problems (n= 28) | 0
  Change at Month 3: Deterioration (n= 27) | 6
  Change at Month 3: No Change (n= 27) | 9
  Change at Month 3: Improvement (n= 27) | 12
  Change at Month 6: Deterioration (n= 28) | 6
  Change at Month 6: No Change (n= 28) | 12
  Change at Month 6: Improvement (n= 28) | 10
  Change at Month 9: Deterioration (n= 28) | 6
  Change at Month 9: No Change (n= 28) | 12
  Change at Month 9: Improvement (n= 28) | 10
  Change at Month 12: Deterioration (n= 28) | 5
  Change at Month 12: No Change (n= 28) | 12
  Change at Month 12: Improvement (n= 28) | 11
  Change at Month 15: Deterioration (n= 27) | 6
  Change at Month 15: No Change (n= 27) | 10
  Change at Month 15: Improvement (n= 27) | 11
  Change at Month 18: Deterioration (n= 24) | 6
  Change at Month 18: No Change (n= 24) | 6
  Change at Month 18: Improvement (n= 24) | 12
  Change at EOT: Deterioration (n= 28) | 6
  Change at EOT: No Change (n= 28) | 9
  Change at EOT: Improvement (n= 28) | 13

12. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Urgency Scale (PPUS) at Months 3,6,9,12,15,18, and End of Treatment
Description: PPUS: self-administered, single-item, questionnaire that measured the participant's perception of urinary urgency. It was sensitive to changes in perceptions of urinary urgency over time. Score of 0 (usually not able to hold urine), 1 (usually able to hold urine [without leaking] until reaching toilet if go to toilet immediately), or 2 (usually able to finish what he/she was doing before going to toilet [without leaking]). Change = observation minus baseline. Deterioration: negative difference of scores; improvement: increase of 1 or more points in difference of scores, relative to baseline.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
Participants
  Baseline: Score 0, Unable to hold urine (n= 28) | 3
  Baseline: Score 1, Able to hold urine (n= 28) | 12
  Baseline:Score 2,Able to finish ongoing task(n=28) | 13
  Change at Month 3: Deterioration (n= 27) | 5
  Change at Month 3: No Change (n= 27) | 17
  Change at Month 3: Improvement (n= 27) | 5
  Change at Month 6: Deterioration (n= 28) | 9
  Change at Month 6: No Change (n= 28) | 13
  Change at Month 6: Improvement (n= 28) | 6
  Change at Month 9: Deterioration (n= 28) | 7
  Change at Month 9: No Change (n= 28) | 19
  Change at Month 9: Improvement (n= 28) | 2
  Change at Month 12: Deterioration (n= 28) | 7
  Change at Month 12: No Change (n= 28) | 17
  Change at Month 12: Improvement (n= 28) | 4
  Change at Month 15: Deterioration (n= 27) | 5
  Change at Month 15: No Change (n= 27) | 19
  Change at Month 15: Improvement (n= 27) | 3
  Change at Month 18: Deterioration (n= 24) | 6
  Change at Month 18: No Change (n= 24) | 12
  Change at Month 18: Improvement (n= 24) | 6
  Change at EOT: Deterioration (n= 28) | 6
  Change at EOT: No Change (n= 28) | 16
  Change at EOT: Improvement (n= 28) | 6

13. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
units on a scale
  Baseline (n= 28) | 35.54 (20.41)
  Month 3 (n= 27) | 33.29 (22.05)
  Month 6 (n= 28) | 32.95 (23.44)
  Month 9 (n= 28) | 33.93 (21.88)
  Month 12 (n= 28) | 29.55 (21.45)
  Month 15 (n= 27) | 31.30 (24.99)
  Month 18 (n= 24) | 31.46 (23.77)
  End of Treatment (n= 28) | 32.59 (23.98)

14. Secondary Outcome: Health Related Quality of Life (HRQL) Domain and Total Score of Overactive Bladder Questionnaire (OAB-q)
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Questions 9 to 33 constitute HRQL, includes domains: concern, coping, sleep, and social function. HRQL domain and total raw score derived as sum of scores. Transformed score range 0 to 100 (Total HRQL or domain) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicative of better HRQL.
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (Week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
units on a scale
  Coping Domain: Baseline (n= 28) | 77.77 (19.69)
  Coping Domain: Month 3 (n= 27) | 78.28 (21.17)
  Coping Domain: Month 6 (n= 28) | 77.14 (21.22)
  Coping Domain: Month 9 (n= 28) | 79.55 (20.67)
  Coping Domain: Month 12 (n= 28) | 76.70 (21.78)
  Coping Domain: Month 15 (n= 27) | 74.54 (23.47)
  Coping Domain: Month 18 (n= 24) | 79.69 (18.61)
  Coping Domain: End of Treatment (n= 28) | 79.29 (18.14)
  Concern Domain: Baseline (n= 28) | 71.04 (18.09)
  Concern Domain: Month 3 (n= 27) | 72.80 (23.20)
  Concern Domain: Month 6 (n= 28) | 70.51 (18.10)
  Concern Domain: Month 9 (n= 28) | 74.49 (19.53)
  Concern Domain: Month 12 (n= 28) | 71.33 (19.73)
  Concern Domain: Month 15 (n= 27) | 69.63 (23.79)
  Concern Domain: Month 18 (n= 24) | 72.50 (21.56)
  Concern Domain: End of Treatment (n= 28) | 72.35 (21.28)
  Sleep Domain: Baseline (n= 28) | 71.00 (19.74)
  Sleep Domain: Month 3 (n= 27) | 73.93 (20.04)
  Sleep Domain: Month 6 (n= 28) | 73.86 (16.85)
  Sleep Domain: Month 9 (n= 28) | 77.04 (19.93)
  Sleep Domain: Month 12 (n= 28) | 74.71 (19.08)
  Sleep Domain: Month 15 (n= 27) | 73.93 (21.89)
  Sleep Domain: Month 18 (n= 24) | 74.33 (21.62)
  Sleep Domain: End of Treatment (n= 28) | 73.57 (21.12)
  Social Interaction Domain: Baseline (n= 28) | 90.57 (10.45)
  Social Interaction Domain: Month 3 (n= 27) | 88.26 (17.25)
  Social Interaction Domain: Month 6 (n= 28) | 87.25 (12.21)
  Social Interaction Domain: Month 9 (n= 28) | 87.11 (15.59)
  Social Interaction Domain: Month 12 (n= 28) | 84.82 (13.42)
  Social Interaction Domain: Month 15 (n= 27) | 84.41 (18.19)
  Social Interaction Domain: Month 18 (n= 24) | 86.79 (17.26)
  Social Interaction Domain: End of Treatment (n=28) | 86.25 (16.69)
  Total: Baseline (n= 28) | 77.09 (16.08)
  Total: Month 3 (n= 27) | 77.87 (19.77)
  Total: Month 6 (n= 28) | 76.65 (16.84)
  Total: Month 9 (n= 28) | 79.14 (18.33)
  Total: Month 12 (n= 28) | 76.42 (18.23)
  Total: Month 15 (n= 27) | 75.01 (21.37)
  Total: Month 18 (n= 24) | 78.02 (18.79)
  Total: End of Treatment (n= 28) | 77.59 (18.32)

15. Secondary Outcome: Number of Participants With Response to Overactive Bladder Satisfaction Questionnaire (OAB-s) (Questions 5, 9, 10a-10d, and 11a-11b)
Description: OAB-s assessed OAB medication expectations, daily life with OAB, and satisfaction with OAB medication. Question (Q) 5 evaluates OAB medication expectations (exceeds/meets or does not meet expectation). Q9 to 11 assessed satisfaction with OAB medication's ability to allow reaching bathroom without urine loss (Q9), decrease: sudden urgencies to urinate (Q10a), urine loss due to urgency (Q10b), waking up at night to urinate (Q10c) and urination during day (Q10d), and improve control of urine loss (Q11a) and need to urinate (Q11b). Q9 to 11 were answered as 'very satisfied', 'somewhat satisfied', 'neither dissatisfied nor satisfied', 'somewhat dissatisfied', and 'very dissatisfied'. The results for Q9 to 11 are reported as "satisfied" (participants who answered 'very satisfied' or 'somewhat satisfied' for all 7 questions) or "not satisfied" (participants who answered 'neither dissatisfied nor satisfied' or 'somewhat dissatisfied' or 'very dissatisfied' for all 7 questions).
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18, End of Treatment (EOT) (Week 82)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
participants
  Baseline, Q5: Exceeding/meeting expectations(n=26) | 22
  Baseline, Q5: Does not meet expectations (n= 26) | 4
  Month 3, Q5: Exceeding/meeting expectations(n=27) | 22
  Month 3, Q5: Does not meet expectations (n= 27) | 5
  Month 6, Q5: Exceeding/meeting expectations(n=28) | 25
  Month 6, Q5: Does not meet expectations (n= 28) | 3
  Month 9, Q5: Exceeding/meeting expectations(n=28) | 25
  Month 9, Q5: Does not meet expectations (n= 28) | 3
  Month 12, Q5: Exceeding/meeting expectations(n=28) | 24
  Month 12, Q5: Does not meet expectations (n= 28) | 4
  Month 15, Q5: Exceeding/meeting expectations(n=27) | 23
  Month 15, Q5: Does not meet expectations (n= 27) | 4
  Month 18, Q5: Exceeding/meeting expectations(n=24) | 19
  Month 18, Q5: Does not meet expectations (n= 24) | 5
  EOT, Q5: Exceeding/meeting expectations(n=28) | 23
  EOT, Q5: Does not meet expectations (n= 28) | 5
  Baseline; Q9, 10a-10d, 11a-11b: Satisfied (n=27) | 19
  Baseline; Q9,10a-10d,11a-11b: Not Satisfied (n=27) | 8
  Month 3; Q9, 10a-10d, 11a-11b: Satisfied (n=26) | 17
  Month 3; Q9,10a-10d,11a-11b: Not Satisfied (n=26) | 9
  Month 6; Q9, 10a-10d, 11a-11b: Satisfied (n=27) | 15
  Month 6; Q9,10a-10d,11a-11b: Not Satisfied (n=27) | 12
  Month 9; Q9, 10a-10d, 11a-11b: Satisfied (n=27) | 16
  Month 9; Q9,10a-10d,11a-11b: Not Satisfied (n=27) | 11
  Month 12; Q9, 10a-10d, 11a-11b: Satisfied (n=27) | 16
  Month 12; Q9,10a-10d,11a-11b: Not Satisfied (n=27) | 11
  Month 15; Q9, 10a-10d, 11a-11b: Satisfied (n=26) | 17
  Month 15; Q9,10a-10d,11a-11b: Not Satisfied (n=26) | 9
  Month 18; Q9, 10a-10d, 11a-11b: Satisfied (n=24) | 16
  Month 18; Q9,10a-10d,11a-11b: Not Satisfied (n=24) | 8
  EOT; Q9, 10a-10d, 11a-11b: Satisfied (n=27) | 18
  EOT; Q9,10a-10d,11a-11b: Not Satisfied (n=27) | 9

16. Secondary Outcome: King's Health Questionnaire (KHQ) Domain Scores
Description: KHQ: self-administered questionnaire contained 21 questions scored in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy, and severity of urinary symptoms). Each domain score ranged: 0-100, where 0=best outcome/response and 100=worst outcome/response.
Time Frame: Baseline, End of Treatment (EOT) (Week 82)
Population: Full analysis set (FAS): included all enrolled participants who had taken at least one dose of study treatment during the study and completed at least one micturition diary. 'n' signifies participants who were evaluable for this measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine
Number analyzed (Participants) | 28
units on a scale
  General Health Perception: Baseline (n=28) | 43.75 (21.11)
  General Health Perception: EOT (n=20) | 38.75 (23.61)
  Incontinence Impact: Baseline (n=27) | 50.62 (23.33)
  Incontinence Impact: EOT (n=20) | 41.67 (26.21)
  Role Limitations: Baseline (n=27) | 31.48 (27.09)
  Role Limitations: EOT (n=20) | 35.00 (30.06)
  Physical Limitations: Baseline (n=27) | 37.04 (30.43)
  Physical Limitations: EOT (n=20) | 34.17 (25.64)
  Social Limitations: Baseline (n=27) | 13.99 (24.19)
  Social Limitations: EOT (n=20) | 20.56 (24.52)
  Personal Relationships: Baseline (n=11) | 1.52 (5.03)
  Personal Relationships: EOT (n=10) | 11.67 (19.33)
  Emotions: Baseline (n=27) | 35.80 (25.66)
  Emotions: EOT (n=20) | 32.78 (22.65)
  Sleep/Energy: Baseline (n=27) | 34.57 (23.08)
  Sleep/Energy: EOT (n=20) | 35.00 (22.88)
  Severity of Urinary Symptoms: Baseline (n=27) | 44.69 (21.86)
  Severity of Urinary Symptoms: EOT (n=20) | 42.33 (21.44)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (N=31)
Epilepsy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine (N=31)
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Blood glucose decreased (Investigations) | 1
Depression (Psychiatric disorders) | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the small sample size and that this is a single country study (Portugal) the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.